CLINICAL TRIAL: NCT01317901
Title: A Phase 1 Study of TRU-016 in Combination With Rituximab and Bendamustine in Subjects With Relapsed Indolent Lymphoma
Brief Title: A Study of TRU-016 in Combination With Rituximab and Bendamustine in Subjects With Relapsed Indolent Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aptevo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16011
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: B-cell Small Lymphocytic Lymphoma Recurrent
Keywords: follicular lymphoma; small lymphocytic lymphoma; marginal zone lymphoma; non-Hodgkin's lymphoma; indolent lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Non-Hodgkin | interventions — TRU 016; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TRU-016+bendamustine+rituximab (Experimental): Two dose levels (10 and 20 mg/kg) of TRU 016 combined with rituximab 375 mg/m2 and bendamustine 90 mg/m2 were evaluated during up to 6 cycles (28 days each). TRU-016 was administered by intravenous (IV) infusion on Days 1 and 15 of each cycle. Rituximab was administered by IV infusion on Day 2 of each cycle. Bendamustine was administered by IV infusion on Days 1 and 2 of each cycle. Subjects received study treatment for up to 6 cycles.
  Interventions: Drug: TRU-016; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: TRU-016 — 100 mg TRU-016 lyophilized solution for infusion at 10 or 20 mg/kg (or 6 mg/kg, if necessary) on Days 1 and 15 of each 28 day cycle
  Other Names: otlertuzumab
Drug: Bendamustine — Bendamustine by IV administration on Days 1 and 2 of each 28 day cycle.
  Other Names: Treanda
Drug: Rituximab — Rituximab by IV administration at 375 mg/m^2 on Day 2 of each 28 day cycle.
  Other Names: rituxan

SUMMARY:
This was a Phase 1 multicenter study of bendamustine, rituximab and TRU-016 (BRT) in subjects with relapsed indolent B-cell lymphoma. This was a multiple-dose escalation study to determine the maximum-tolerated dose (MTD) of TRU-016 given in combination with rituximab and bendamustine and to determine a safe dosing regimen for the combination in up to 12 subjects with relapsed indolent lymphoma.

The originally planned Phase 2 portion, an open-label, randomized study to evaluate the efficacy of BRT compared with BR, was not conducted.

DETAILED DESCRIPTION:
This study was planned to be conducted in 2 parts: a Phase 1b component designed to determine a safe dosing regimen, and a Phase 2 component designed to evaluate the efficacy of BRT compared to BR in subjects with relapsed indolent lymphoma. The Phase 2 component was not conducted.

This was an open-label, non randomized, multiple-dose escalation study to determine the MTD of BRT and to determine a safe dosing regimen for the combination in subjects with relapsed indolent lymphoma.

The study consisted of a screening period lasting up to 21 days, a treatment period lasting up to 6 cycles (28 days each), and a 60-day follow-up period. Up to 12 subjects (2 cohorts of 6 subjects each) were planned for enrollment. Two dose levels (10 and 20 mg/kg) of TRU-016 combined with rituximab 375 mg/m2 and bendamustine 90 mg/m2 were evaluated during up to 6 cycles (28 days each). TRU-016 was administered by intravenous (IV) infusion on Days 1 and 15 of each cycle. Rituximab was administered by IV infusion on Day 2 of each cycle. Bendamustine was administered by IV infusion on Days 1 and 2 of each cycle. Subjects received study treatment for up to 6 cycles.

ELIGIBILITY:
Inclusion Criteria

1. Age 18 years or older
2. Histologically confirmed diagnosis of indolent non-Hodgkin's B-cell lymphoma (ie, follicular lymphoma, small lymphocytic lymphoma, and marginal zone lymphoma) that has relapsed (relapsed is defined as confirmed progressive disease (PD) after receiving the most recent prior therapy, or failure to achieve at least a partial response (PR) while receiving the most recent prior therapy)
3. At least one prior line of therapy for indolent lymphoma
4. Bi-dimensionally measurable disease with at least one lesion measuring >=1.5 cm in a single dimension
5. Eastern Cooperative Oncology Group (ECOG) performance status of <= 2
6. Creatinine clearance of >40 mL/min as calculated by the

Cockcroft-Gault method as follows:

(140 - age) * (weight in kg [* 0.85 if female] / 72 * serum creatinine level) 7. Adequate hepatic function, indicated as follows:

* aspartate aminotransferase (AST) of <2.5 x upper limit of normal (ULN)
* alanine aminotransferase (ALT) of <2.5 x ULN
* total bilirubin of <= 1.5 x ULN 8. Absolute neutrophil count (ANC) >=1000/mm3 (1000/µL) 9. Platelet count >= 100,000/mm3 10. Female subjects of child-bearing potential and male subjects must use an acceptable form of birth control for the duration of their study participation and for 6 months after completing study drug dosing; acceptable forms of birth control, unless dictated otherwise by local regulatory authorities 11. For women of childbearing potential, a negative serum pregnancy test result obtained during the screening period and a negative urine pregnancy test result within 24 hours before first administration of study drug 12. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information

Exclusion Criteria

1. Diagnosis of grade 3b follicular lymphoma or transformed lymphoma of any grade
2. Previously received TRU-016
3. Prior treatment with rituximab if subject discontinued rituximab due to unresolved toxicity
4. Refractory to bendamustine, defined as follows:

   * progression within 6 months of last dose of bendamustine
   * failed to achieve at least a PR while receiving bendamustine
   * discontinued bendamustine due to toxicity
   * received bendamustine within 6 months prior to first dose of study drug
5. Received chemotherapy, radiotherapy, or immunotherapy including investigational agents within 28 days prior to the first dose of study drug
6. Received therapeutic corticosteroids at doses equivalent to >10 mg prednisone per day for longer than 5 days within 14 days prior to the first dose of study drug, except if needed as a pre-medication
7. Received filgrastim or equivalent within 14 days prior to screening (ie, collection of samples for laboratory tests) or pegfilgrastim within 28 days prior to screening (ie, collection of samples for laboratory tests)
8. Prior allogeneic bone marrow transplant
9. Prior autologous bone marrow transplant within 12 months prior to the first dose of study drug
10. Received blood or platelet infusion within 7 days prior to screening (ie, collection of samples for laboratory tests)
11. Previous or concurrent additional malignancy except non-invasive, non-melanomatous skin cancer or in situ carcinoma of the cervix, or other solid tumors if the subject has been disease-free for a minimum of 2 years prior to the first dose of study drug
12. Known central nervous system or leptomeningeal lymphoma
13. Any significant concurrent medical diseases or conditions, including but not limited to the following:

    * Clinically significant pulmonary dysfunction requiring oxygen therapy
    * An active infection (viral, bacterial, or fungal) requiring systemic therapy; subjects receiving prophylactic therapy are eligible
14. Known allergy to mannitol
15. History of positive serology for human immunodeficiency virus (HIV)
16. Positive serology for hepatitis B (surface antigen or core antibody) Note: If a positive test result for hepatitis B core antibody is due to immunoglobulin treatment, the subject may be enrolled if the hepatitis B viral deoxyribonucleic acid (DNA) is negative.
17. Positive serology for hepatitis C
18. Pregnant or breastfeeding
19. Other severe, acute, or chronic medical or psychiatric condition, laboratory abnormality, or difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration or may interfere with safety
20. Any condition that, in the investigator's opinion, makes the subject unsuitable for study participation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-05; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Stromatt, MD, Study Director — Aptevo Therapeutics
Locations (6):
- United States (6):
  - Site Reference ID/Investigator# 61543, Birmingham, Alabama
  - Site Reference ID/Investigator# 61542, Augusta, Georgia
  - Site Reference ID/Investigator# 61523, Omaha, Nebraska
  - Site Reference ID/Investigator# 61522, Hackensack, New Jersey
  - Site Reference ID/Investigator# 61544, Chapel Hill, North Carolina
  - Site Reference ID/Investigator# 61524, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gopal AK, Tarantolo SR, Bellam N, Green DJ, Griffin M, Feldman T, Mato AR, Eisenfeld AJ, Stromatt SC, Goy A. Phase 1b study of otlertuzumab (TRU-016), an anti-CD37 monospecific ADAPTIR therapeutic protein, in combination with rituximab and bendamustine in relapsed indolent lymphoma patients. Invest New Drugs. 2014 Dec;32(6):1213-25. doi: 10.1007/s10637-014-0125-2. Epub 2014 Jun 15. PMID 24927856

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve adult patients, 6 in each dose group, were enrolled at 4 hospitals between May and October 2011.
Groups:
- 10 mg/kg TRU-016+Bendamustine+Rituximab; 20 mg/kg TRU-016+Bendamustine+Rituximab: TRU-016: 100 mg TRU-016 lyophilized solution for infusion at 10 mg/kg (or 6 mg/kg, if necessary) on Days 1 and 15 of each 28 day cycle Rituximab: 375 mg/m^2 rituximab was administered by IV infusion on Day 2 of each cycle.
  Bendamustine: 90 mg/m^2 bendamustine was administered by IV infusion on Days 1 and 2 of each cycle.
Period: Overall Study
Arm/Group | 10 mg/kg TRU-016+Bendamustine+Rituximab | 20 mg/kg TRU-016+Bendamustine+Rituximab
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRU-016 (10 mg/kg) +Bendamustine+Rituximab | TRU-016 (20 mg/kg) +Bendamustine+Rituximab | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (4.76) | 64.3 (10.61) | 60.8 (8.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 5 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
β2-microglobulin [Mean (Standard Deviation); unit: MG/l] | 2.4 (1.3) | 2.9 (1.9) | 2.6 (1.5)
Sum of product diameters [Mean (Standard Deviation); unit: cm2] | 40.9 (26.5) | 35.0 (32.6) | 37.9 (28.5)
Time since first diagnosis of primary cancer [Mean (Standard Deviation); unit: years] | 3.2 (2.8) | 6.0 (4.7) | 4.6 (4.0)
Direct Anti-globulin Test [Number; unit: participants]
  Positive | 0 | 0 | 0
  Negative | 6 | 5 | 11
  unknown | 0 | 1 | 1
Staging at diagnosis [Number; unit: participants]
  Stage 1 | 1 | 0 | 1
  Stage 2 | 1 | 1 | 2
  Stage 3 | 1 | 2 | 3
  Stage 4 | 2 | 3 | 5
  Not done | 1 | 0 | 1
FLIPI [Number; unit: participants] — Follicular Lymphoma International Prognostic Index
  participants
    Low risk (0-1 points) | 3 | 3 | 6
    Intermediate risk (2 points) | 3 | 1 | 4
    Highrisk (3-5 points) | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Response was assessed by the investigator on the basis of clinical, radiological, and pathological (i.e., bone marrow) criteria, using the IWG criteria (Cheson et al 2007). A CR is a complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy. A PR is at least a 50% decrease in sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses, no increase should be observed in the size of other nodes, liver or spleen, and no new sites of disease should be observed.
Time Frame: Day 15 and Day 28 of even-numbered cycles
Population: All treated subjects
Measure: Number; unit: participants
Groups:
- TRU-016 (10 mg/kg) + Bendamustine + Rituximab: 10 mg/kg of TRU 016 combined with rituximab 375 mg/m^2 and bendamustine 90 mg/m^2 were evaluated during up to 6 cycles (28 days each). TRU-016 was administered by intravenous (IV) infusion on Days 1 and 15 of each cycle. Rituximab was administered by IV infusion on Day 2 of each cycle. Bendamustine was administered by IV infusion on Days 1 and 2 of each cycle. Subjects received study treatment for up to 6 cycles.
  TRU-016: 100 mg TRU-016 lyophilized solution for infusion at 10 or 20 mg/kg (or 6 mg/kg, if necessary) on Days 1 and 15 of each 28 day cycle
  Bendamustine: Bendamustine by IV administration on Days 1 and 2 of each 28 day cycle.
  Rituximab: Rituximab by IV administration at 375 mg/m^2 on Day 2 of each 28 day cycle.
- 20 mg/kg of TRU 016 + Bendamustine + Rituximab: 20 mg/kg of TRU 016 combined with rituximab 375 mg/m^2 and bendamustine 90 mg/m^2 were evaluated during up to 6 cycles (28 days each). TRU-016 was administered by intravenous (IV) infusion on Days 1 and 15 of each cycle. Rituximab was administered by IV infusion on Day 2 of each cycle. Bendamustine was administered by IV infusion on Days 1 and 2 of each cycle. Subjects received study treatment for up to 6 cycles.
Arm/Group | TRU-016 (10 mg/kg) + Bendamustine + Rituximab | 20 mg/kg of TRU 016 + Bendamustine + Rituximab
Number analyzed (Participants) | 6 | 6
participants
  Complete Response | 3 | 2
  Partial Response | 1 | 4
  Stable disease | 1 | 0
  Relapsed/progressive disease | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: After initiation of study medications (TRU-016, rituximab, or bendamustine), all adverse events (AEs) and serious adverse events (SAEs) regardless of attribution were collected until 60 days following the last administration of study treatment or initiation of new therapy, whichever was earlier.
Groups:
- TRU-016 (10 mg/kg): TRU-016 (10 mg/kg) + bendamustine + rituximab
- TRU-016 (20 mg/kg): TRU-016 (20 mg/kg) + bendamustine + rituximab
Arm/Group | TRU-016 (10 mg/kg) | TRU-016 (20 mg/kg)
Serious Adverse Events (participants affected / at risk) | 2/6 | 3/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRU-016 (10 mg/kg) (N=6) | TRU-016 (20 mg/kg) (N=6)
febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
pneumonia (Infections and infestations) | 1 | 1
vestibular disorder (Ear and labyrinth disorders) | 1 | 1
retinal vein occlusion (Eye disorders) | 1 | 1
myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRU-016 (10 mg/kg) (N=6) | TRU-016 (20 mg/kg) (N=6)
neutropenia (Blood and lymphatic system disorders) | 5 | 2
anemia (Blood and lymphatic system disorders) | 2 | 1
thrombocytopenia (Blood and lymphatic system disorders) | 3 | 3
lymphopenia (Blood and lymphatic system disorders) | 1 | 1
febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
vestibular disorder (Ear and labyrinth disorders) | 1 | 1
retinal vein occlusion (Eye disorders) | 1 | 1
nausea (Gastrointestinal disorders) | 3 | 4
abdominal pain (Gastrointestinal disorders) | 3 | 3
diarrhea (Gastrointestinal disorders) | 1 | 2
vomiting (Gastrointestinal disorders) | 1 | 2
constipation (Gastrointestinal disorders) | 0 | 2
dry mouth (Gastrointestinal disorders) | 1 | 0
dyspepsia (Gastrointestinal disorders) | 0 | 1
hemorrhoids (Gastrointestinal disorders) | 1 | 1
fatigue (General disorders) | 3 | 4
chill (General disorders) | 0 | 2
influenza ike illness (General disorders) | 1 | 0
Non-cardiac chest pain (Cardiac disorders) | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
White blood cell count decreased (Investigations) | 3 | 1
Neutrophil count decreased (Investigations) | 3 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Lymphocyte count decreased (Investigations) | 2 | 0
Aspartate aminotransferase (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Immunoglobulins decreased (Investigations) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 2 | 1
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Phlebitis (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No